CLINICAL TRIAL: NCT06674304
Title: Registry Initiative Across Borders for Atrial Fibrillation in Africa
Acronym: RIBATAFRICA-AF
Status: Active, not recruiting | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, RAISSUNI Zainab, Professor of cardiology, Mohammed VI University Hospital
Other Study IDs: Mohammed VI UH Tangier
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation (Prevention of Stroke); ATRIAL FIBRILLATION, Syncope
Keywords: Atrial fibrillation; Registry; Africa; Morocco; antithrombotic treatment
MeSH Terms: conditions — Atrial Fibrillation; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Atrial fibrillation is a penalizing disease in several ways: morbidity and mortality, health costs. Several multicenter registries have been published. Until now, no multicenter registry involving several countries has been carried out in Africa. The goal of RIBAT AF Africa is to fill this gap, by recruting patients from twelve african centers. All the centers are a third level Atrial Fibrillation managment facility centers.

After recruitment , a complete clinical assessment with analysis of comorbidities will be a priority of this registry to try to understand the epidemiological profile of atrial fibrillation in Africa. Then, we will proceed to the temporal classification of atrial fibrillation according to the 2024 ESC recommendations (type and thromboembolic risk in particular.).

After this step, the management will be analyzed with three main axes: management of comorbidities, antithrombotic treatment, rhythm and frequency control. Some therapeutic techniques such as ablation of atrial fibrillation were discussed without much detail because many countries do not yet have access to these expensive techniques.

A six-month evaluation is necessary to judge above all the applicability of the measures accessible in all countries and in particular anticoagulant treatment.

All these data will be recorded anonymously and electronically. Each country can have access to its own data anytime. The statistical analysis will be carried out by a team within the University Hospital of Tangier , as well as all IT logistics. This team will also organize electronic monitoring and underlying all abnomalities in CRF.

DETAILED DESCRIPTION:
I. Rational

Atrial fibrillation is a penalizing disease in several ways: morbidity and mortality, health costs. Several multicenter registries have been published. Until now, no multicenter registry involving several countries has been carried out. The goal of RIBAT AF Africa is to fill this gap.

II. Study objectives

* To understand the epidemiological profile of atrial fibrillation in Africa,
* to describe the management of atrial fibrillation in Morocco
* to proceed to the temporal classification of atrial fibrillation according to the 2024 ESC recommendations (type and thromboembolic risk in particular.),
* to analyze and describe the management of comorbidities,
* to describe the antithrombotic treatment,
* to study the association between heart failure with preserved ejection fraction and FA
* to analyze the rhythm and frequency control.
* to describe the imaging features in FA

III. Study timeline

A six-month evaluation is necessary to judge above all the applicability of the measures accessible in all countries and in particular anticoagulant treatment. The data collection's start estimation is planned for October 2024. Result will be available in October 2025.

IV. Project description

1. Study design

   This is a multicentric, prospective and observational study, that will be held simultaneously in 13 african countries. The Moroccan center represented by the Mohammed VI university hospital is the coordinating center as well as the principal investigator (PI) center for this study.
2. Population

   About 3000 patients will be included in the study according to the following criteria:

   Inclusion criteria
   * Patients aged ≥ 18 years old
   * Patients with a documented history of AF for any length of time before enrolment or AF first diagnosed at enrolment visit/hospitalization
   * Patients previously diagnosed with AF must have at least one documented visit or hospitalization for AF (or AF-related complications) within the last 12 months before enrolment Exclusion criteria
   * No formal diagnosis of AF in medical records
   * Only atrial flutter or other atrial tachycardia diagnosed
   * Participation in a clinical trial (but participation in another registry is allowed)

   For the sampling procedures, all patients who meet the inclusion criteria, and followed for management in the study centers, will be included exhaustively until the needed number of subjects is reached.
3. Procedure

   1. Investigators

      The 'RIBAT-AFRICA-FA' registry brings together 13 investigating centers in 13 countries; Benin, Cameroun, Egypt, Ethiopia, Gabon, Ivory Coast, Kenya, Mauritania, Morocco, Mali, Niger, Senegal and Tunisia. Each investigating center is located in a university hospital and chaired by a professor of cardiology. In Morocco, the cardiology department of the Mohammed VI University Hospital is the coordinating centre and main investigator. It also coordinates the inclusion of patients in several private cardiology practices in order to ensure that the data is representative of the whole of Morocco.
   2. Data collection

      A Case Report Form (CRF) has been developed by the Moroccan Society of Cardiology, and will be used to collect anamnestic, clinical, exploratory and therapeutic data, as well as six-month outcomes (see appendix).

      For each patient included in this study, the CRF will be completed at inclusion, throughout the initial management period and after six months of treatment.
   3. Data managment The RIBAT-AFRICA-FA registry will be managed by the Epidemiology and Public Health team and the IT team at CHU Mohammed VI of Tangiers.

   For data collection, an electronic CRF (eCRF) has been created on the CHU Mohammed VI of Tanger's RedCap application. For each investigating center, a private account was created and communicated. In addition, a training session on the use of the eCRF was organized for all investigators.

   Throughout the study period, monitoring and data quality management will be carried out by the epidemiology team at CHU Mohammed VI de Tanger.

   Supervision and coordination of the registry is the responsibility of the Head of Cardiology at Tangier University Hospital.
4. Statistical Analysis

Statistical analysis will be performed using IBM SPSS version 25 software. Descriptive data for continuous variables will be presented as means/standard deviation or Median/IQR according to the normality of the distributions, while qualitative variables will be presented as percentages with 95% confidence intervals. Chi-square, Student's t-test or ANOVA will be used within the limits of their respective validity conditions, and where appropriate, non-parametric tests will be used. Multivariate analyses may be indicated, in which case logistic regression and/or the Cox model may be used depending on the model.

V. Ethical Considerations

1. Funding The project is sponsored by the Moroccan laboratory Afric-Phar, which is facilitating and taking charge of all logistical aspects of project implementation, including coordination between the investigating centers.

   The sponsor will not have access to the data circuit from collection to statistical analysis and publication.
2. Conflit of interest no conflicts of interest to declare.
3. Patient's information Patients will have access to a detailed information sheet before their inclusion. Each investigator will explain in a very satisfactory manner the objectives of the study as well as its contribution for improving medical knowledge concerning FA. No additional risk is incurred by the patients included, in particular each patient has the right to refuse participation without this refusal impacting the normal course of the care process.
4. Consent information Informed consent Will be obtained from each patient before its inclusion.
5. Other ethical considerations The data collected as part of this project will be processed in accordance with all standards of good practice and confidentiality preservation.

The data will be stored on a secure server owned by the University Hospital Center (CHU).

No additional paraclinical investigations will be conducted outside of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old
* Patients with a documented history of AF for any length of time before enrolment or AF first diagnosed at enrolment visit/hospitalization
* Patients previously diagnosed with AF must have at least one documented visit or hospitalization for AF (or AF-related complications) within the last 12 months before enrolment

Exclusion Criteria:

* No formal diagnosis of AF in medical records
* Only atrial flutter or other atrial tachycardia diagnosed
* Participation in a clinical trial (but participation in another registry is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 3000 patients will be included in the study according to the following criteria:
  Inclusion criteria
  * Patients aged ≥ 18 years old
  * Patients with a documented history of AF for any length of time before enrolment or AF first diagnosed at enrolment visit/hospitalization
  * Patients previously diagnosed with AF must have at least one documented visit or hospitalization for AF (or AF-related complications) within the last 12 months before enrolment Exclusion criteria
  * No formal diagnosis of AF in medical records
  * Only atrial flutter or other atrial tachycardia diagnosed
  * Participation in a clinical trial (but participation in another registry is allowed)
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Arial fibrillation complications under treatment | Six month follow up
  After inclusion, the investigators carry out a six-month follow-up for the patients. During this prospective follow-up period, the primary judgment criterion that must be documented by the investigators is the occurrence of a complication linked to AF or its medical management. The main complications to be looked for are :
  1. Death
  2. Non fatal stroke or systemic embolic event
  3. Non fatal haemorrhagic event
  4. Drug side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed VI University Hospital of Tangier, Tangier, Tangier, Morocco

IPD SHARING:
Plan to Share IPD: Undecided